CLINICAL TRIAL: NCT01307982
Title: Comparative Anti-Reflux Procedures in Neurologically Impaired Children
Acronym: CARPNIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Raj Srivastava, Dr. Raj Srivastava, MD, MPH, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00043616
Record Dates: First submitted 2011-02-18; First posted 2011-03-03 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Gastroesophageal Reflux; Nervous System Diseases; Fundoplication; Enteral Nutrition
Keywords: Gastroesophageal Reflux; Nervous System Diseases; Fundoplication; Enteral Nutrition
MeSH Terms: conditions — Gastroesophageal Reflux; Nervous System Diseases | interventions — Fundoplication; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fundoplication (Active Comparator): During fundoplication surgery, the upper curve of the stomach (the fundus) is wrapped around the esophagus and sewn into place so that the lower portion of the esophagus passes through a small tunnel of stomach muscle. This surgery strengthens the valve between the esophagus and stomach (lower esophageal sphincter), which stops acid from backing up into the esophagus as easily.
  Interventions: Procedure: Fundoplication
- Gastrojejunal (GJ) feeding tube (Active Comparator): Gastrojejunal (GJ) tube placement is an image guided technique in which a special soft feeding catheter is placed through an existing hole in the stomach (gastrostomy) into the small bowel (jejunum).
  Interventions: Procedure: Gastrojejunal (GJ) feeding tube

INTERVENTIONS:
Procedure: Fundoplication — During fundoplication surgery, the upper curve of the stomach (the fundus) is wrapped around the esophagus and sewn into place so that the lower portion of the esophagus passes through a small tunnel of stomach muscle. This surgery strengthens the valve between the esophagus and stomach (lower esophageal sphincter), which stops acid from backing up into the esophagus as easily.
  Other Names: Nissen Fundoplication
  Arms: Fundoplication
Procedure: Gastrojejunal (GJ) feeding tube — Gastrojejunal (GJ) tube placement is an image guided technique in which a special soft feeding catheter is placed through an existing hole in the stomach (gastrostomy) into the small bowel (jejunum).
  Other Names: GJ tube
  Arms: Gastrojejunal (GJ) feeding tube

SUMMARY:
This trial is a randomized controlled trial of two standard anti-reflux procedures, Nissen fundoplication versus gastrojejunal feeding tubes (GJ tubes), in children and adolescents with functional and intellectual impairment who have gastrostomy feeding tubes and medically refractory or severe gastroesophageal reflux disease (GERD). This is a pilot study to establish feasibility before initiating a multi-centered study.

ELIGIBILITY:
Inclusion Criteria:

* patient is between 6 months and 18 years of age; AND
* patient has functional impairment classified by either gross motor functional classification of 3, 4 or 5 OR impaired function in walking, crawling/standing, rolling/sitting, arm use, hand use, ability to hold head up; AND
* patient has a gastrostomy; AND
* patient has intolerance of feedings or other complications attributed to GERD as defined below; AND
* patient has a positive GERD diagnostic evaluation as define below:

  * GERD diagnostic evaluation will include the following investigations;

    * endoscopy and biopsy for visual assessment and histology of the esophageal mucosa
    * pH study and/or multichannel intraluminal impedance (MII) probe to detect and quantify gastroesophageal reflux
  * GER demonstrated by:

    * Reflux Esophagitis: Endoscopic appearance of mucosal breaks in the distal esophagus with or without pathologist diagnosis based on one or more biopsy histologic features of: inflammatory cellular infiltrate, basal cell hyperplasia, elongation of the vascular papillae AND no infectious microorganisms and < 15 eosinophils per high power field; OR
    * pH OR pH/multichannel intraluminal impedance(MII) probe evidence of pathologic GER:

      * pH probe: acid reflux index > 7 % OR
      * pH/MII reflux symptom-associated acid or non-acid volume associated reflux events;
  * Upper GI will only be used to determine normal anatomy; AND
* patient has either medically refractory GERD or severe GERD as defined below:

  * Medically refractory GERD - GERD that has not responded to 12 weeks of treatment with a proton pump inhibitor (PPI) (and verified gastric pH > 4) and/or trial of continuous intragastric feedings and has one of the following complications:

    * Esophagitis: Endoscopic appearance of mucosal breaks in the distal esophagus with or without pathologist diagnosis based on one or more biopsy histologic features of: inflammatory cellular infiltrate, basal cell hyperplasia, elongation of the vascular papillae
    * Failure to thrive: diminishing weight percentile for age or weight for age z-score sustained over 6 months.
    * Pneumonia consistent with aspiration,
    * Acute life threatening event,
  * Severe GERD - at least one severe complication of GERD and patient cannot safely tolerate a trial of medical management due to one of the following life-threatening complications:

    * aspiration pneumonia,
    * acute life threatening event (ALTE),
    * complete loss of airway protection (absent cough/gag) AND,
* Upper GI barium contrast study for anatomy; AND
* Barium pharyngeal swallow study or modified barium swallow study or Flexible Endoscopic Evaluation of Swallowing (FEES) in past year; AND
* the parent or legal guardian speaks English or Spanish (the only two languages in which the instruments are standardized)

Exclusion Criteria:

* Upper GI findings that would mandate a fundoplication including: hiatal hernia, esophageal stricture, Barret's esophagus; OR
* Upper GI findings show uncorrected distal gastrointestinal obstruction including: gastric outlet obstruction, duodenal obstruction, malrotation; OR
* Upper GI demonstrates structural foregut abnormalities that preclude a fundoplication including: microgastria, short esophagus, high anesthetic risk; OR
* Diagnosis or history of congenital diaphragmatic hernia, esophageal atresia, chronic intestinal pseudoobstruction; OR
* Endoscopy and biopsy demonstrates esophagitis from causes other than GER including: eosinophilic esophagitis, candida esophagitis, viral esophagitis); OR
* Rapidly changing or indeterminate neurological including either a deteriorating neurological condition such as rapid loss of developmental milestones or improving, such as rapid recovery following severe neurological insult; OR
* Patient has unacceptable general anesthetic risk; OR
* A previous Nissen fundoplication; OR
* Feeds delivered by GJ/NJ at the time of enrollment occurring for greater than 3 months.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
GERD-related hospitalization and ED visits | 12 months
  Parental interviews and chart reviews will be used to record all health care encounters. Each encounter will be classified as either GERD-related or not. GERD-related hospitalizations and ED visits will be further classified as; diagnostic testing, procedural problems, likely aspiration pneumonia (AP or bacterial pneumonia), respiratory distress of other etiology, or death from any cause.

SECONDARY OUTCOMES:
Health Related Quality of Life | 12 months
  These are a series of surveys about the child and caregiver's health related quality of life.
Total length of stay | 12 months
  This is the length of stay for each hospitalization and ED visit.
Complications from treatment | 12 months
  This will be monitored with hospitalizations (primary outcome)
Complications from failure of treatment | 12 months
  This will be monitored with hospitalizations (primary outcome), and will include things such as repeat procedure for fundoplication arm, ongoing need for GERD medications, and treatment cross-over.
Mortality | 12 months
  Any cause captured at 28 days and 12 months post procedure. Procedure related deaths will also be captured.
Costs related to hospital, ED, outpatient, and home-health care | 12 months
  This will be abstracted from hospital administrative database.
Nutritional outcomes | 12 months
  Nutritional outcomes will be measured through anthropomorphic measurements including:
  * weight for age z-score
  * tibial length
  * triceps and subscapular skinfold thickness
Other outpatient health care | 12 months
  This will include primary care provider, neurology, gastroenterology, surgery, physiotherapy, etc.
Symptom control | 12 months
  We will ask parents/caregivers to evaluate their childs symptoms and severity.
Parental Goals of either treatment for GERD | 12 months
  We will ask parents/caregivers their goals for treatment and evaluate if they have been met.
Physician Goals of either treatment for GERD | 12 months
  We will ask physicians their goals for treatment and evaluate if they have been met.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Srivastava, MD, MPH, Principal Investigator — University of Utah
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States